CLINICAL TRIAL: NCT05204121
Title: Phase Ib, Single-Center, Randomized Study of Safety, Tolerability and Pharmacokinetics of Elpida in Healthy HIV-Uninfected Volunteers
Brief Title: Phase Ib Study of Safety, Tolerability and Pharmacokinetics of Elpida Once Weekly in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HIV-VM1500-09
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — elsulfavirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Elpida 40 mg once weekly (Experimental): elsulfavirine 40mg orally once weekly for 8 weeks
  Interventions: Drug: Elpida
- Elpida 80 mg once weekly (Experimental): elsulfavirine 80mg orally once weekly for 8 weeks
  Interventions: Drug: Elpida
- Elpida 160 mg once weekly (Experimental): elsulfavirine 160mg orally once weekly for 8 weeks
  Interventions: Drug: Elpida

INTERVENTIONS:
Drug: Elpida — elsulfavirine, capsules
  Other Names: elsulfavirine; VM-1500; VM1500

SUMMARY:
A randomized once weekly dose for 8 weeks, study in Healthy HIV-Uninfected Volunteers. Each of 3 parallel groups (40 mg, 80 mg and 160mg) enrolls 12 subjects.

DETAILED DESCRIPTION:
The study aims to assess safety, tolerability and PK of once weekly administration of Elpida in different doses.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 55 years;
2. Verified diagnosis "healthy" according to medical history, physical examination, assessment of vital signs, electrocardiography (ECG), investigations performed in the last 14 days prior to the first administration of IP;
3. Body mass index (BMI) from 18.5 kg/m2 to 30 kg/m2 (inclusive), bodyweight of 50 kg or higher;
4. Negative result of alcohol and drug tests;
5. Women must be in postmenopause for at least 2 years, be surgically sterile or use two reliable methods of contraception from the day of screening and until 3 months after the last dose;
6. Men must use two reliable methods of contraception* from the day of screening and until 3 months after the last dose;
7. Ability to understand the meaning of the study and any risks associated with participation. Ability to interact with the investigator, participate and comply with the requirements of the study throughout its duration;
8. Willingness to sign written consent to participate in the study after reading Informed Consent Form with the opportunity to discuss any questions with the investigator (and/or his/her representative).

Exclusion Criteria:

1. Participation in more than one group of investigational therapy;
2. Past or present diseases of the cardiovascular, bronchopulmonary, neuroendocrine, musculoskeletal systems, as well as diseases of the gastrointestinal tract, liver, kidneys, blood that may interfere with achievement of objectives of this study or affect the safety of a volunteer;
3. The values of laboratory and instrumental parameters, beyond the limit of normal ;
4. Past or present diseases or pathologies, including surgical interventions in the gastrointestinal tract that, in the opinion of the Investigator, may affect the absorption, distribution, metabolism or excretion of the investigational product;
5. A systolic pressure of less than 90 mm Hg or greater than 130 mm Hg; diastolic pressure of less than 60 mm Hg or greater than 85 mm Hg; pulse rate of less than 60 bpm or greater than 90 bpm (at screening);
6. Deviations detected during 12-lead ECG, or QT/QTc interval > 450 milliseconds (ms) for men and > 470 ms for women;
7. Administration of any drugs n, including over-the-counter products, herbal, food, dietary or vitamin supplements 14 days before the first administration of the investigational product;
8. Administration of the following drugs for 28 days prior to screening: corticosteroids (any route of administration); IP that inhibit the activity of cytochrome P450 3A4 (CYP3A4; for example, ritonavir and other drugs for human immunodeficiency virus (HIV), ketoconazole, itraconazole, or similar azole antifungals and macrolide antibiotics such as erythromycin), or the use of any drugs with a significant likely effect on functions of organs (for example, barbiturates, omeprazole, cimetidine);
9. Hepatitis B (HBsAg), antibodies to hepatitis C and HIV, a positive test for syphilis;
10. Positive pregnancy test (for women);
11. Acute infectious diseases less than 4 weeks before screening;
12. Unstable sleeping hours (for example, night shift, sleep disorders, insomnia, jet lag, etc.);
13. Signs of alcohol or drug addiction; intake of alcohol or drugs 4 days prior to screening and during the study; smoking cigarettes 3 months prior to screening and during the study; positive drug and/or alcohol test;
14. Complicated allergic history (including intolerance to medication, including hypersensitivity to the active substance/excipients of the investigational drug) and food allergy;
15. Blood/plasma donation (450 mL of blood or plasma or more) less than 2 months before screening;
16. Participation in another clinical study or administration of any investigational products less than 3 months before screening;
17. Any other concomitant medical or significant mental conditions that render a volunteer unsuitable for participation in the clinical study;
18. A volunteer who is considered for enrollment in the study is an employee of the study site or company of the Sponsor or a member of an employee's family

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs and SAEs | 77 days
  Incidence of AEs and SAEs

SECONDARY OUTCOMES:
elsulfavirine plasma concentration | 77 days
  elsulfavirine plasma concentration
VM1500A plasma concentration | 77 days
  active metabolite plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Elena Smolyarchuk, MD, PhD, Principal Investigator — Sechenov First Moscow State Medical University
Locations (1):
- Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided